CLINICAL TRIAL: NCT03519802
Title: Evaluation of Cognitive Function in a Suicidal Crisis and Interest to Achieve a MoCA Test in Acute Situations
Brief Title: Evaluation of Cognitive Function in a Suicidal Crisis
Acronym: CocaCS
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2015_84; 2016-A00881-50 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-04-26; First posted 2018-05-09 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2020-09

CONDITIONS: Suicide
Keywords: Cognitive functions; MoCA test
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aftermath of suicide is devastating, being the cause of 800 000 deaths every year worldwide. In France, suicide still causes about 10 000 deaths per year and the number of suicide attempts (SA) is estimated between 170 000 and 200 000 per year (InVS).

It is often thought that a suicidal crisis is only related to depression, as it actually is a far more complex phenomenon. A suicidal crisis can occur on various grounds like psychiatric disorders but also contextual events or somatic diseases and it has been hypothesized that suicidal ideas or inclinations could have a common and independent cognitive origin

ELIGIBILITY:
Inclusion Criteria:

* Normal or corrected vision
* Having understood the information not and having signed the form of consent
* Being hospitalized for suicidal ideas (Score with inclusion at the level of Beck > 3) or after a suicide attempt of less than one week.

Exclusion criteria:

* Pregnant woman and/or nursing
* Diagnosed irrational pathology
* Known proven intellectual deficiency
* Patient whose physical or mental status does not allow to pass the tests of the study
* Being under supervision or trusteeship or private of freedom or in emergency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients hospitalized for less than a week and presenting with a suicidal crisis
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Rate of patients having a score in MoCA test strictly under 26 | at inclusion

SECONDARY OUTCOMES:
Variation in MoCA test scores between before (V1) and after hospitalization (V2) | an average at 3 months after inclusion
Variation in scores to the subtests between between before (V1) and after hospitalization (V2) | an average at 3 months after inclusion
Rate of patients having lower subtests scores than the standards | an average at 3 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Vincent JARDON, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU,Hôpital Fontan, Lille, France

IPD SHARING:
Plan to Share IPD: No